CLINICAL TRIAL: NCT02418572
Title: Transdermal Testosterone Gel for Poor Ovarian Responders. A Multicenter Double-blind Placebo Controlled Randomized Trial
Brief Title: Testosterone TRANSdermal Gel for Poor Ovarian Responders Trial
Acronym: T-TRANSPORT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Having reached the sample size described for the interim analysis and having seen the post-interim results, the sponsor has decided to stop the trial due to futility.
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Nikolaos Polyzos, Principal Investigator, Fundacion Dexeus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014.TTRANSPORT; 2014-001835-35 (EudraCT Number)
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Infertility; Poor Ovarian Response
MeSH Terms: conditions — Infertility | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transdermal testosterone gel (Experimental): Patients will receive once daily application of 0.55 gr TTG (Testosterone gel 1%; Laboratories Besins International,Paris,France) with a 5.5 mg/d nominal delivery rate of testosterone starting from day 1 or 2 of the following menstrual cycle, for approximately 65 days.
  Pituitary down-regulation will be induced by daily injections of 0.1mg triptorelin started on day 21 of the next cycle following enrollment in the study, up to and including the day of hCG administration.
  After 2 weeks of down-regulation, daily SC injections of HP-hMG (Menopur®) (300 IU/day) will be administered up to the day of hCG administration.
  Ovulation triggering will be induced with 250μg rhCG (Ovidrelle®) followed by oocyte pick-up ~36 hours later and ICSI. A maximum of 2 embryos, following each center's national criteria of single embryo transfer, will be transferred 3 days later.
  Luteal phase support with be performed with progesterone tablets ( Utrogestan®) (200mg x3, intravaginally).
  Interventions: Drug: Testosterone gel
- Placebo transdermal gel (Placebo Comparator): Patients will receive once daily application of 0.55 gr identical placebo gel starting from day 1 or 2 of the following menstrual cycle, for approximately 65 days.
  Pituitary down-regulation will be induced by daily injections of 0.1mg triptorelin started on day 21 of the next cycle following enrollment in the study, up to and including the day of hCG administration.
  After 2 weeks of down-regulation, daily SC injections of HP-hMG (Menopur®) (300 IU/day) will be administered up to the day of hCG administration.
  Ovulation triggering will be induced with 250μg rhCG (Ovidrelle®) followed by oocyte pick-up ~36 hours later and ICSI. A maximum of 2 embryos, following each center's national criteria of single embryo transfer, will be transferred 3 days later.
  Luteal phase support with be performed with progesterone tablets ( Utrogestan®) (200mg x3, intravaginally).
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: Testosterone gel — Patients will receive once daily application of 0.55 gr testosterone gel-TTG (GROUP A) (Testosterone gel 1%; Laboratories Besins International, Paris, France) with a 5.5 mg/d nominal delivery rate of testosterone starting from day 1 or 2 of the following menstrual cycle, for approximately 65 days.
  The application will be administered in the morning by the patient onto clean dry healthy skin over external surface of the thighs. The gel will be simply spread on the skin gently as a thin layer.
  TTG will start on the day of enrollment and will continue until patients' menstruation (28-30 days). Daily administration of TTG or placebo will continue for 35 days (21days until the initial of downregulation with triptorelin and for 14 more days until the initiation of ovarian stimulation with HP-hMG). Ovarian stimulation will commence the day after last testosterone gel application. (GROUP A)
  Other Names: Androgel 1% 0.55 gr / day
  Arms: Transdermal testosterone gel
Drug: Placebo gel — Patients will receive once daily application of 0.55 gr of placebo gel from day 1 or 2 of the following menstrual cycle, for approximately 65 days.
  The application will be administered in the morning by the patient onto clean dry healthy skin over external surface of the thighs. The gel will be simply spread on the skin gently as a thin layer.
  Placebo gel will start on the day of enrollment and will continue until patients' menstruation (28-30 days). Daily administration of placebo gel will continue for 35 days (21 days until the initial of downregulation with triptorelin and for 14 more days until the initiation of ovarian stimulation with HP-hMG
  Arms: Placebo transdermal gel

SUMMARY:
Previous work indicates that 2 months androgen pre-treatment may equip preantral follicles with more FSH receptors and increase the cohort of follicles surviving to the recruitable antral stage. In this regard it may result in an increase in the oocyte yield and the reproductive outcome in women with poor ovarian response. These findings provide a strong rationale for a definitive large RCT. The TTRANSPORT study will include 400 women with poor ovarian response randomized to receive pre-treatment with transdermal testosterone gel or placebo in order to provide conclusive evidence regarding the superiority or not of transdermal testosterone pre-treatment for the management of poor ovarian responders fulfilling the Bologna criteria.

DETAILED DESCRIPTION:
Studies in primates showed that treatment with testosterone increased the number of growing follicles, lead to proliferation of granulosa and theca cells, while finally reduced the apoptosis of granulosa cells (Vendola et al., 1999; Weil et al., 1999). These studies further suggest that androgens may have a specific action in pre-antral and small antral follicles, prior to serving as substrate for estradiol synthesis in larger follicles and in this regard influence the responsiveness of the ovaries to gonadotropins and amplify the effects of FSH on the ovary.

Despite the available evidence, only 3 small RCTs evaluated the effect of transdermal testosterone on infertile patients with poor ovarian response to stimulation. A pooled analysis of these studies demonstrated a benefit in clinical and ongoing pregnancy rates for testosterone pre-treated patients (González-Comadran et al., 2012). However, two of these trials were considerably small, whereas all of them restricted testosterone administration between 5 and 21 days prior ovarian stimulation. Evidence from basic research and early trials suggest that androgens should be administered for at least 2 months before initiation of ovarian stimulation (Casson PR, 2000), in order affect preantral follicles and equip them with more FSH receptors in an attempt to have a larger cohort of follicles surviving to the recruitable antral stage.

Taking into account the promising results from recently conducted small RCTS, the investigators decided to perform a double blind placebo controlled randomized controlled trial, with adequate sample size, in order to test the effect of administration of transdermal testosterone in poor ovarian responders fulfilling the Bologna criteria, for 2 months prior ovarian stimulation in a long agonist protocol. The daily dose of transdermal testosterone gel (TTG) will be 0.55gr (5.5mg testosterone/day). The specific dose was selected based on previous pharmacokinetic studies in women according to which daily application of 5 mg of transdermal testosterone cream (Fooladi, 2014) or TTG (Singh et al. 2006, Nathorst-Böös et al., 2005) is likely to restore fT levels to the premenopausal reference range. Although no side effects had been described after pre-treatment with higher doses of 12.5mg TTG for 21 days in a previous randomized controlled trial (Kim et al., 2011), it is likely that higher doses will result in supraphysiological TT and fT levels. Therefore the dose of 0.55gr TTG (5.5mg testosterone/day) has been selected for the T-TRANSPORT trial since this will restore TT and fT levels to levels above and within the upper normal reference range.

ELIGIBILITY:
Inclusion Criteria:

Patients participating in the TTRANSPORT study will be women who are considered poor ovarian responders according to the "Bologna criteria" (Ferraretti et al., 2011).

Subjects must fulfil the following criteria to be included in the study:

1. All subjects must sign the Informed consent documents prior to screening evaluations.
2. Age: between 18-43 years old.
3. One of the features below:

Infertile female <40 years old with i. ≤ 3 oocytes in a previous cycle and AFC <7 OR ii. ovarian surgery/chemotherapy and AFC<7 OR iii. ≤ 3 oocytes in at least 2 previous cycles with ≥300IU gonadotropins

Infertile female ≥40 years old with i. ≤ 3 oocytes in a previous cycle OR ii. AFC <7. Patients will be randomized according to different age groups (<36, 36-39 and ≥40 years old).

Exclusion Criteria:

1. Perimenopausal women with amenorrhea not having a regular cycle
2. Basal FSH >20 IU/l
3. Uterine malformations
4. Recent history of any current untreated endocrine abnormality
5. Unilateral or bilateral hydrosalpinx (visible on USS, unless clipped)
6. Contraindications for the use of gonadotropins
7. Recent history of severe disease requiring regular treatment
8. Use of androgens during the last 3 months
9. Patients with SHBG values <20nmol/L or >160nmol/L
10. Azoospermia (sperm derived through FNA or TESE)

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 290 (Actual)
Dates: Start 2015-04; Primary Completion 2023-12 (Actual); Study Completion 2024-02 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | 7 weeks of gestation
  The presence of intrauterine gestational sac with an embryonic pole demonstrating cardiac activity at 7 weeks of gestation

SECONDARY OUTCOMES:
Ongoing pregnancy | 9-10 weeks of gestation
  The presence of intrauterine gestational sac with an embryonic pole demonstrating cardiac activity at 9-10 weeks of gestation.
Biochemical pregnancy | 2 weeks after embryo transfer
  Positive pregnancy test 2 weeks after embryo transfer
Number of oocytes retrieved | 9 -20 days from initiation of ovarian stimulation
  The outcome will be evaluated on the day of oocyte retrieval
Number of MII oocytes retrieved | 9 -20 days from initiation of ovarian stimulation
  The outcome will be evaluated on the day of oocyte retrieval
Cycle cancellation due to poor ovarian response | 10 days after initiation of daily injections of HP-hMG
  On stimulation day 10 (visit 8) the cycle will be cancelled in case of no follicular or monofollicular development
Number of cycles reaching the stage of embryo transfer | 9 -20 days from initiation of ovarian stimulation
  The outcome will be evaluated 3 days after oocyte retrieval
Number and quality of embryos | Day of embryo transfer (9 -20 days from initiation of ovarian stimulation)
  The outcome will be evaluated 3 days after oocyte retrieval
Number of cycles with frozen supernumerary embryos | 9 -20 days from initiation of ovarian stimulation
  The outcome will be evaluated 5 days after oocyte retrieval or 2-6 days after embryo transfer in case of an embryo transfer

OTHER OUTCOMES:
Adverse events | Up to 70 days from treatment start date
  Any adverse event related with testosterone administration must be reported in Adverse Event Report Form

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos P Polyzos, MD PhD, Principal Investigator — Fundacion Dexeus
Locations (10):
- Universitair Ziekenhuis Brussel, Brussels, Belgium
- Denmark (2):
  - Fertility Clinic Rigshospitalet, Copenhagen
  - The Fertility Clinic, Skive Regional Hospital, Skive, Denmark, Skive
- Spain (6):
  - Hospital Universitario Quiron Dexeus, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Monteprincipe, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospìtal Universitario HM Puerta del Sur, Madrid
  - Quiron Madrid Hospital, Madrid
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Background] Casson PR, Lindsay MS, Pisarska MD, Carson SA, Buster JE. Dehydroepiandrosterone supplementation augments ovarian stimulation in poor responders: a case series. Hum Reprod. 2000 Oct;15(10):2129-32. doi: 10.1093/humrep/15.10.2129. PMID 11006185
- [Background] Gonzalez-Comadran M, Duran M, Sola I, Fabregues F, Carreras R, Checa MA. Effects of transdermal testosterone in poor responders undergoing IVF: systematic review and meta-analysis. Reprod Biomed Online. 2012 Nov;25(5):450-9. doi: 10.1016/j.rbmo.2012.07.011. Epub 2012 Jul 26. PMID 22999555
- [Background] Vendola K, Zhou J, Wang J, Famuyiwa OA, Bievre M, Bondy CA. Androgens promote oocyte insulin-like growth factor I expression and initiation of follicle development in the primate ovary. Biol Reprod. 1999 Aug;61(2):353-7. doi: 10.1095/biolreprod61.2.353. PMID 10411511
- [Background] Weil S, Vendola K, Zhou J, Bondy CA. Androgen and follicle-stimulating hormone interactions in primate ovarian follicle development. J Clin Endocrinol Metab. 1999 Aug;84(8):2951-6. doi: 10.1210/jcem.84.8.5929. PMID 10443703
- [Background] Kim CH, Howles CM, Lee HA. The effect of transdermal testosterone gel pretreatment on controlled ovarian stimulation and IVF outcome in low responders. Fertil Steril. 2011 Feb;95(2):679-83. doi: 10.1016/j.fertnstert.2010.07.1077. PMID 20801436
- [Background] Singh AB, Lee ML, Sinha-Hikim I, Kushnir M, Meikle W, Rockwood A, Afework S, Bhasin S. Pharmacokinetics of a testosterone gel in healthy postmenopausal women. J Clin Endocrinol Metab. 2006 Jan;91(1):136-44. doi: 10.1210/jc.2005-1640. Epub 2005 Nov 1. PMID 16263817
- [Background] Nathorst-Boos J, Jarkander-Rolff M, Carlstrom K, Floter A, von Schoultz B. Percutaneous administration of testosterone gel in postmenopausal women--a pharmacological study. Gynecol Endocrinol. 2005 May;20(5):243-8. doi: 10.1080/09513590500097283. PMID 16019368
- [Background] Fooladi E, Reuter SE, Bell RJ, Robinson PJ, Davis SR. Pharmacokinetics of a transdermal testosterone cream in healthy postmenopausal women. Menopause. 2015 Jan;22(1):44-9. doi: 10.1097/GME.0000000000000259. PMID 24845394
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Derived] Leathersich SJ, Davis SR, Garcia Martinez S, Blockeel C, Martinez F, Gosalvez A, Humaidan P, de la Fuente L, Fabregues F, Pinborg A, Stoop D, Polyzos NP. The impact of transdermal testosterone treatment on quality of life in women with diminished ovarian reserve: secondary analysis of a randomized controlled trial. Hum Reprod. 2025 Dec 29:deaf233. doi: 10.1093/humrep/deaf233. Online ahead of print. PMID 41461161